CLINICAL TRIAL: NCT03488238
Title: Correlation of Changes in PaO2 and ORi in Adult Patients
Status: Completed | Type: Interventional
Sponsor: Masimo Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: FLEM0007
Record Dates: First submitted 2018-03-29; First posted 2018-04-04 (Actual); Results first posted 2021-09-20 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-08

CONDITIONS: Hyperoxia
MeSH Terms: conditions — Hyperoxia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- ORi sensor (Experimental): All subjects are enrolled in the test group and receive an ORi sensor during their scheduled, general surgery procedure
  Interventions: Device: ORi sensor

INTERVENTIONS:
Device: ORi sensor — Noninvasive pulse oximeter sensor that is placed on the finger for measurement of ORi

SUMMARY:
The Oxygen Reserve Index (ORi) is a reference that could help clinicians with their assessments of normoxic and hyperoxic states by scaling the measured absorption information between 0.00 and 1.00. An ORi of 0.00 corresponds to PaO2 values of 100mmHg and below and an ORi of 1.00 corresponds to PaO2 values of 200mmHg and above. This is a prospective, non-blinded, non-randomized study of the Oxygen Reserve Index (ORi) in a clinical setting. It is designed to evaluate the correlations with ORi and changes in PaO2 and the potential use of ORi as an early warning of impending arterial oxygen desaturation.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* ASA physical status III or IV
* Scheduled for an elective surgical procedure requiring endotracheal intubation and the use of an arterial pressure monitoring catheter placed prior to induction of general anesthesia

Exclusion Criteria:

* Age less than 18 years
* Adults unable to give primary consent
* Pregnancy
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-09-19 (Actual); Study Completion 2018-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UC Davis, Sacramento, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ORi Sensor
Started | 31
Completed | 29
Not Completed | 2
Not completed — Equipment malfunction | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | ORi Sensor
Number analyzed (Participants) | 29
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 29

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity for Changes in ORi Values as Compared to Corresponding Changes in PaO2 Values.
Description: ORi is an index value without a unit and ORi does not directly measure PaO2. Therefore, sensitivity is calculated to evaluate changes in ORi relative to the changes in PaO2.
Time Frame: Less than 30 mins
Population: 1 subject was excluded as investigator reported unreliable data.
Measure: Number; unit: percentage of true positives
Arm/Group | ORi Sensor
Number analyzed (Participants) | 28
percentage of true positives | 100

2. Primary Outcome: Specificity for Changes in ORi Values as Compared to Corresponding Changes in PaO2 Values.
Description: ORi is an index value without a unit and ORi does not directly measure PaO2. Therefore specificity is calculated to evaluate changes in ORi relative to the changes in PaO2.
Time Frame: Less than 30 mins
Population: 1 subject was excluded as investigator reported unreliable data.
Measure: Number; unit: percentage of true negatives
Arm/Group | ORi Sensor
Number analyzed (Participants) | 28
percentage of true negatives | 94.38

3. Primary Outcome: Concordance for Changes in ORi Values as Compared to Corresponding Changes in PaO2 Values.
Description: ORi is an index value without a unit and ORi does not directly measure PaO2. Therefore concordance is calculated to evaluate changes in ORi relative to the changes in PaO2.
Time Frame: Less than 30 minutes
Population: 1 subject was excluded as investigator reported unreliable data.
Measure: Number; unit: percentage of accuracy
Arm/Group | ORi Sensor
Number analyzed (Participants) | 28
percentage of accuracy | 95.05

ADVERSE EVENTS:
Time Frame: Less than 30 min
Arm/Group | ORi Sensor
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 1/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ORi Sensor (N=29)
Hypotension (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/38/NCT03488238/Prot_SAP_000.pdf